CLINICAL TRIAL: NCT06526988
Title: Implementation and Interaction of Clinician And Patient-facing Tools Aiming to Intensify Neurohormonal Medicines for Heart Failure With Reduced Ejection Fraction: I-I-CAPTAIN-HF
Brief Title: Implementation and Interaction of Clinician And Patient-facing Tools Aiming to Intensify Neurohormonal Medicines for Heart Failure
Acronym: IICAPTAIN-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Yale University (Other); Northwestern University (Other); University of Utah (Other); Sutter Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 24-1449; BPS-2023C1-31460 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart failure; Patient-centered care; Clinical decision support; Guideline-directed medical therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Cluster-randomization will occur at the clinician level, where the clinician is randomized to 1 of 4 study arms (usual care, EPIC-HF only, PROMPT-HF only, both). Randomization will be stratified at the site level. Patient assignment follows clinician randomization.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (No Intervention): Patients will receive care as usual.
- EPIC-HF Patient-facing Tool (Experimental): Patients will receive the patient engagement video and HeartMeds Guide checklist electronically about 2-7 days and 0-1 days prior to their next clinic appointment after enrollment.
  Interventions: Behavioral: EPIC-HF Patient-facing Tool
- PROMPT-HF Clinician-facing Alert (Experimental): Clinicians will receive tailored electronic health record (EHR) alerts recommending guideline-directed medical therapy (GDMT) in eligible patients with HFrEF during outpatient visits.
  Interventions: Behavioral: PROMPT-HF Clinician-facing Alert
- Both (EPIC-HF and PROMPT-HF Interventions) (Experimental): Patients will receive the patient engagement video and HeartMeds Guide checklist electronically about 2-7 days and 0-1 days prior to their next clinic appointment after enrollment, and clinicians will receive tailored electronic health record (EHR) alerts recommending guideline-directed medical therapy (GDMT) in eligible patients with HFrEF during outpatient visits.
  Interventions: Behavioral: EPIC-HF Patient-facing Tool; Behavioral: PROMPT-HF Clinician-facing Alert

INTERVENTIONS:
Behavioral: EPIC-HF Patient-facing Tool — A brief, animated video designed to engage and activate patients around their HFrEF medication prescribing sent prior to routine cardiology clinic visit, accompanied by a one-page HeartMeds Guide checklist.
  Arms: Both (EPIC-HF and PROMPT-HF Interventions); EPIC-HF Patient-facing Tool
Behavioral: PROMPT-HF Clinician-facing Alert — A best practice alert will appear for each eligible patient upon opening of the order entry screen in the patient's medical record. This alerts the provider of the presence of HFrEF, notes the patient's current LVEF and current evidence-based medications, and gives access to an order set with recommended evidence-based, guideline-recommended, and FDA- approved therapies for patients with HFrEF. Providers will also have access to a link to best available guideline recommended information regarding treatment of heart failure to allow further education if desired by the provider. The alerts will also clearly state the expected monitoring and follow-up required for prescriptions of these medications.
  Arms: Both (EPIC-HF and PROMPT-HF Interventions); PROMPT-HF Clinician-facing Alert

SUMMARY:
An increasing number of guideline-directed medical therapies (GDMT) have been developed for patients with chronic heart failure with reduced ejection fraction (HFrEF). When used in combination at recommended doses, patients often experience significant improvements in cardiac function, quality of life, and survival.1,2 However, GDMT underuse occurs for the vast majority of patients with HFrEF. Two recent trials demonstrated improved GDMT prescribing during a clinic visit, each using automated delivery of a patient-centered decision support tool to promote a proactive and holistic approach to prescribing: EPIC-HF (NCT03334188) tested a brief video and checklist document sent to patients just prior to a clinic visit encouraging them to work with their clinicians to make at least 1 positive change to their GDMT; PROMPT-HF (NCT05433220) tested tailored electronic health record (EHR) alerts for GDMT intensification delivered to clinicians during clinic visits. The current I-I-CAPTAIN-HF study aims to broadly implement and test the EPIC-HF patient-facing and PROMPT-HF clinician-facing tools for HFrEF medication intensification at 5 health systems around the country through a pragmatic cluster-randomized implementation-effectiveness trial. This will occur through an initial phase of adaptation of the 2 tools at each health system. Once ready, the 2 tools will be tested using a 2x2 randomization at the clinician-level. In parallel, formal assessment of the implementation of EPIC-HF and PROMPT-HF will work to understand the most effective means of intervention design and delivery, as well as adaptations due to contextual factors to optimize use.

DETAILED DESCRIPTION:
I-I-CAPTAIN-HF is a multi-site, type-2 hybrid implementation-effectiveness trial conducted at 5 sites: the University of Colorado (central site), Yale University, Northwestern University, University of Utah, and Sutter Health.

Aim 1. Implement the EPIC-HF and PROMPT-HF interventions at 5 health systems through participatory work with a multi-level team using the PRISM framework to guide the delivery of a host of implementation strategies that respect mandatory aspects of the interventions (function) and explore adaptations (form) to maximize equitable reach, broad adoption, fidelity of implementation, and long-term maintenance.

* Hypothesis 1A: Standard EHR logic (in Epic) can be created for HFrEF identification and automated delivery of both interventions, followed by tailoring to individual system EHR infrastructure.
* Hypothesis 1B: Challenges around automated intervention delivery can be identified, solutions developed, and processes shared for optimal integration into the local clinic environment.
* Hypothesis 1C: Issues of equity-digital access, language, out-of-pocket cost, social determinants of health-can be addressed by intervention and delivery adaptations, respecting uniqueness of recipients.

The initial phase of I-I-CAPTAIN-HF explores a host of implementation strategies that will take the existing EPIC-HF and PROMPT-HF interventions and optimize their ability to be implemented widely while retaining tool fidelity. Current versions of EPIC-HF and PROMPT-HF were tested in single sites under research conditions that have led to barriers to wider uptake. In Aim 1, the investigators and study team will 1) form an External Advisory Committee, 2) apply PRISM domains to define mandatory functions of the interventions, 3) engage site partners to define form adaptations using the iPRISM web tool to assess context, 4) vet adaptable forms to consider fidelity to function, 5) decide final forms for each site, and 6) pilot local versions of each interventions using EHR technical testing to ensure feasibility, usability, and acceptability. The tools will be implemented and automated within each EHR and used as standard of care for all eligible patients.

Prior to conclusion of Aim 1, all sites will pilot test their site-based implementation approach to assess feasibility, usability, and user acceptability before widespread implementation in Aim 2. This process will conclude with interviews with team members to assess the fidelity to the intervention, as well as gather data on adaptations to the intervention by each site. These interviews will be conducted by the central site (University of Colorado) study team and occur with those involved at each site with implementing the interventions and could include site-principal investigators and/or co-investigators, IT leadership or analysts.

Aim 2. Test the effectiveness, as well as the interaction, of the EPIC-HF and PROMPT-HF interventions to improve GDMT prescribing from before to after the clinic visit among 2000 patients at 5 health systems using a 2x2 factorial design randomized at the clinician-level.

* Hypothesis 2A - Effectiveness: Both EPIC-HF and PROMPT-HF will improve GDMT intensification.
* Hypothesis 2B - Interaction: Patient- and clinician-facing tools may work better when used in combination.

Cluster-randomization will occur at the clinician level, where the clinician is randomized to 1 of 4 study arms (usual care, EPIC-HF only, PROMPT-HF only, both). Randomization will be stratified at the site level. Patient assignment follows clinician randomization.

Following processes developed in Aim 1, each site will deliver the assigned intervention(s) to patients and clinicians as per randomization. Those clinicians randomized to intervention(s) will have the intervention delivered to the clinician themselves (PROMPT-HF) and/or their patient (EPIC-HF) prior to the patient's scheduled routine clinic appointment. The interventions will be implemented as standard of care across those in the intervention arms and occur for all eligible patients.

Patient-level data will be collected through the patients' EHRs.

Aim 3. Evaluate ongoing implementation of EPIC-HF and PROMPT-HF using Practical, Robust Implementation and Sustainability Model (PRISM) to understand the most effective means of intervention design and delivery, as well as adaptations due to contextual factors.

• Hypothesis 3: Understanding key mandatory elements and tailored adaptations to the interventions and their delivery will maximize equitable impact across implementation outcomes (reach), increase uptake by the clinics and their clinicians (adoption), ease appropriate deployment (implementation and adaptations), and lead to sustained use after the clinical trial (maintenance).

Implementation of EPIC-HF and PROMPT-HF will be explored using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) outcomes from the PRISM framework to understand the most effective means of sustainable delivery.

Reach: Investigators will attempt to characterize the proportion and representativeness of eligible patients who receive the intervention. Representativeness will be assessed by comparing participants who opt in versus those who opt out based on demographic/clinical indicators.

Effectiveness: Assessed in Aim 2, above.

Adoption: The absolute number, proportion, and representativeness of settings and intervention agents (clinicians) who are willing to initiate a program will be assessed. Effectively, adoption should be 100% at the site level since all programs who were approached have agreed to participate. Data will be collected on adoption at the clinician level, where each clinician can enroll or decline at study start, and then adopt or ignore PROMPT-HF CDS during study conduct. Clinicians' attitudes towards the new approach will be explored using clinician surveys measured before and after the trial.

Implementation: The investigators will assess the extent to which the intervention is implemented as intended (fidelity) and adaptations made. With a mixed methods evaluation, the experiences of EPIC-HF and PROMPT-HF and their combination will be explored.

Maintenance: The study team will systematically collect data on local decisions regarding maintenance and will also assess staff recommendations for sustainment.

ELIGIBILITY:
Inclusion Criteria:

Clinician:

* Clinician (MD, PA, NP) who practices in cardiology outpatient clinics
* Regularly sees patients with left ventricular ejection fraction (EF) </=40%, where their panel of patients over the last year included at least 25 patients with heart failure with reduced ejection fraction (HFrEF)

Patient:

* Age > 18 years
* LVEF </=40% on most recent cardiology imaging study
* Has had a routine cardiology outpatient clinic appointment in the previous 12 months
* Not on all 4 pillars of GDMT at optimal doses: (1) beta blockers, (2) angiotensin receptor-neprilysin inhibitor/angiotensin converting enzyme inhibitor/angio-tensin receptor blocker, (3) aldosterone receptor antagonists, (4) sodium-glucose co-transporter

Exclusion Criteria:

Patient:

* Has a left ventricular assist device
* Under evaluation for or listed for transplant (or s/p transplant)
* Glomerular filtration rate (GFR) less than 15
* On IV inotropes
* On hospice care
* Non-English or Non-Spanish speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Intensification of GDMT in patients with Heart Failure with Reduced Ejection Fraction | From pre-clinic visit to 1 day after
  The primary outcome for this trial is the proportion of patients with HFrEF who have an increase in the number of prescribed HFrEF therapies (beta blockers, ACE-I/ARB/ARNI, MRA, SGLT2i) and/or dosing intensification from pre-clinic visit to 1 day after.

SECONDARY OUTCOMES:
Individual drug class changes | 0, 1, 30 days
  Change in the number of prescribed HFrEF therapies and/or dosing intensification for the following: beta blockers, ACE-I/ARB/ARNI, MRA, SGLT2i.
Safety and adverse events | 1-90 days
  Hospitalizations and emergency room visits with diagnosis of hypotension, bradycardia, acute renal failure, hyperkalemia, allergic reaction to medication, urinary tract infection, worsening heart failure, and other.
Patient activation | Day after visit
  In a survey sent to patients, the Patient Assessment of Chronic Illness Care (PACIC) will be collected. This is a patient-level assessment of healthcare that focuses on the receipt of patient-centered care and self-management behaviors. Scores on the PACIC range from 1 to 5, with higher scores indicating patient's perception of greater involvement in self-management and receipt of chronic care counseling. The PACIC sub-domains of 'Patient Activation' and 'Five As' Agree' will be used for this study.
Patient Self efficacy | Day after visit
  In a survey sent to patients, the Decision Self Efficacy Scale will be collected. It measures self-confidence or belief in one's ability in decision making, including shared decision making. A score of 0 means 'extremely low self efficacy' and a score of 100 means 'extremely high self efficacy'.
Clinician attitudes toward patient activation tools and clinical decision support | Baseline, at study completion (about 2.5 years)
  In a survey sent to clinicians, a six-item attitudes measure adapted for EPIC-HF and PROMPT-HF interventions will be collected.
Clinician acceptability and feasibility of interventions | At study completion (about 2.5 years)
  In a survey sent to clinicians, Acceptability of Intervention Measure and Feasibility of Intervention Measure will be collected.
Reach of EPIC-HF intervention | Throughout study period (about 2.5 years)
  Reach of the EPIC-HF intervention will be measured by the proportion and representativeness of eligible patients who receive the intervention. Representativeness will be assessed by comparing participants who opt in versus those who opt out based on demographic/clinical indicators.
Adoption of PROMPT-HF intervention | Throughout study period (about 2.5 years)
  Adoption of the PROMPT-HF intervention will be measured by the proportion and representativeness of eligible clinicians who enroll versus decline.
Implementation of PROMPT-HF and EPIC-HF interventions | Throughout study period (about 2.5 years), day after visit for patient, at study completion (about 2.5 years) for clinician
  In a survey sent to clinicians and patients, questions on their use and opinions of the PROMPT-HF and EPIC-HF interventions will be collected. In a subset of clinicians and patients, qualitative interviews will be conducted to get a more in-depth understanding of implementation.
Maintenance of PROMPT-HF and EPIC-HF interventions | 6 months after primary data collection completion
  Rate of continued use of interventions after study period through interviews with site clinicians and institutional leadership.

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Allen, MD, MHS, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - Sutter Health, Walnut Creek, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Only aggregate participant data will be reported. A de-identified study dataset will be available on a data repository website after study collection and analysis is completed.

REFERENCES:
- [Background] Allen LA, Venechuk G, McIlvennan CK, Page RL 2nd, Knoepke CE, Helmkamp LJ, Khazanie P, Peterson PN, Pierce K, Harger G, Thompson JS, Dow TJ, Richards L, Huang J, Strader JR, Trinkley KE, Kao DP, Magid DJ, Buttrick PM, Matlock DD. An Electronically Delivered Patient-Activation Tool for Intensification of Medications for Chronic Heart Failure With Reduced Ejection Fraction: The EPIC-HF Trial. Circulation. 2021 Feb 2;143(5):427-437. doi: 10.1161/CIRCULATIONAHA.120.051863. Epub 2020 Nov 17. PMID 33201741
- [Background] Venechuk GE, Khazanie P, Page RL 2nd, Knoepke CE, Helmkamp LJ, Peterson PN, Pierce K, Thompson JS, Huang J, Strader JR, Dow TJ, Richards L, Trinkley KE, Kao DP, McIlvennan CK, Magid DJ, Buttrick PM, Matlock DD, Allen LA. An Electronically delivered, Patient-activation tool for Intensification of medications for Chronic Heart Failure with reduced ejection fraction: Rationale and design of the EPIC-HF trial. Am Heart J. 2020 Nov;229:144-155. doi: 10.1016/j.ahj.2020.08.013. Epub 2020 Aug 28. PMID 32866454
- [Background] Swat SA, Helmkamp LJ, Tietbohl C, Thompson JS, Fitzgerald M, McIlvennan CK, Harger G, Ho PM, Ahmad FS, Ahmad T, Buttrick P, Allen LA. Clinical Inertia Among Outpatients With Heart Failure: Application of Treatment Nonintensification Taxonomy to EPIC-HF Trial. JACC Heart Fail. 2023 Nov;11(11):1579-1591. doi: 10.1016/j.jchf.2023.06.022. Epub 2023 Aug 16. PMID 37589610
- [Background] Venechuk G, Allen LA, Thompson JS, Morris MA, Matlock DD, McIlvennan CK, Dickert NW, Tietbohl C. Trust and activation in defining patient-clinician interactions for chronic disease management. Patient Educ Couns. 2023 Jan;106:113-119. doi: 10.1016/j.pec.2022.09.012. Epub 2022 Sep 22. PMID 36167759
- [Background] Ghazi L, Yamamoto Y, Riello RJ, Coronel-Moreno C, Martin M, O'Connor KD, Simonov M, Huang J, Olufade T, McDermott J, Dhar R, Inzucchi SE, Velazquez EJ, Wilson FP, Desai NR, Ahmad T. Electronic Alerts to Improve Heart Failure Therapy in Outpatient Practice: A Cluster Randomized Trial. J Am Coll Cardiol. 2022 Jun 7;79(22):2203-2213. doi: 10.1016/j.jacc.2022.03.338. Epub 2022 Apr 3. PMID 35385798
- [Background] Desai AS, Maclean T, Blood AJ, Bosque-Hamilton J, Dunning J, Fischer C, Fera L, Smith KV, Wagholikar K, Zelle D, Gaziano T, Plutzky J, Scirica B, MacRae CA. Remote Optimization of Guideline-Directed Medical Therapy in Patients With Heart Failure With Reduced Ejection Fraction. JAMA Cardiol. 2020 Dec 1;5(12):1430-1434. doi: 10.1001/jamacardio.2020.3757. PMID 32936209
- [Background] Mebazaa A, Davison B, Chioncel O, Cohen-Solal A, Diaz R, Filippatos G, Metra M, Ponikowski P, Sliwa K, Voors AA, Edwards C, Novosadova M, Takagi K, Damasceno A, Saidu H, Gayat E, Pang PS, Celutkiene J, Cotter G. Safety, tolerability and efficacy of up-titration of guideline-directed medical therapies for acute heart failure (STRONG-HF): a multinational, open-label, randomised, trial. Lancet. 2022 Dec 3;400(10367):1938-1952. doi: 10.1016/S0140-6736(22)02076-1. Epub 2022 Nov 7. PMID 36356631
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Dunlay SM, Killian JM, Roger VL, Schulte PJ, Blecker SB, Savitz ST, Redfield MM. Guideline-Directed Medical Therapy in Newly Diagnosed Heart Failure With Reduced Ejection Fraction in the Community. J Card Fail. 2022 Oct;28(10):1500-1508. doi: 10.1016/j.cardfail.2022.07.047. Epub 2022 Jul 25. PMID 35902033
- [Background] Greene SJ, Butler J, Albert NM, DeVore AD, Sharma PP, Duffy CI, Hill CL, McCague K, Mi X, Patterson JH, Spertus JA, Thomas L, Williams FB, Hernandez AF, Fonarow GC. Medical Therapy for Heart Failure With Reduced Ejection Fraction: The CHAMP-HF Registry. J Am Coll Cardiol. 2018 Jul 24;72(4):351-366. doi: 10.1016/j.jacc.2018.04.070. PMID 30025570
- [Background] Kilsdonk E, Peute LW, Jaspers MW. Factors influencing implementation success of guideline-based clinical decision support systems: A systematic review and gaps analysis. Int J Med Inform. 2017 Feb;98:56-64. doi: 10.1016/j.ijmedinf.2016.12.001. Epub 2016 Dec 5. PMID 28034413